CLINICAL TRIAL: NCT05665036
Title: A Phase 1/2 Open-Label, Sequential Dose-Escalation, Safety, Tolerability and Efficacy Study of SIG-005 in Adult Patients With Mucopolysaccharidoses 1 (MPS-1)
Brief Title: Safety and Efficacy of Encapsulated Allogeneic MPS-1 Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor developing new product
Sponsor: Sigilon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIG-005-121
Record Dates: First submitted 2021-11-03; First posted 2022-12-27 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: MPS I; MPS1-S; MPS1-HS
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SIG-005 (Experimental): SIG-005 is comprised of human native alpha-L-iduronidase enzyme (hIDUA) producing spheres
  Interventions: Combination Product: SIG-005 (hIDUA Producing Spheres)

INTERVENTIONS:
Combination Product: SIG-005 (hIDUA Producing Spheres) — Laparoscopic administration of SIG-005 spheres, an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce hIDUA

SUMMARY:
SIG-005-121 is a FIH, Phase 1/2, multi-centre, open-label, sequential dose-escalating study to assess the safety, tolerability, and preliminary efficacy of SIG-005 in adults with MPS-1. The study will evaluate up to three ascending dose levels of SIG-005 in male and female patients with attenuated MPS-1 (Scheie or Hurler-Scheie), 18 years of age or greater, who received Enzyme Replacement Therapy (ERT) for a minimum of 12 months prior to the study entry. Each cohort will include 3 patients.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Male or female aged 18 or older
* Diagnosis of attenuated MPS-1 (Hurler-Scheie or Scheie)
* Alpha-L-iduronidase enzyme activity level of less than 10% of the lower limit of the normal range
* Prior treatment with ERT
* Willing to transition from ERT to SIG-005
* Female patients of childbearing potential with negative pregnancy test
* Use of highly effective method of contraception if applicable

Exclusion Criteria:

* A diagnosis of severe MPS-1
* Previous haematopoietic stem cell transplantation (HSCT)
* History of elevated total (IgG) anti-IDUA antibody
* Use of assistive respiratory devices
* Unable to walk independently
* History of allergic reaction or anaphylaxis to recombinant hIDUA
* Body mass index (BMI) ≥35
* History of abdominal adhesions, medical history of Crohn's disease, inflammatory bowel disease or any disease that increases the risk of post-operative abdominal adhesions
* Significant underlying disease or comorbidities that are a contraindication for general anaesthesia or laparoscopic procedure
* Pregnant or lactating patients
* Prior administration of a gene therapy product
* Participation in another investigational medicine or device study
* Abnormal laboratory values as defined in the protocol
* Active alcoholism or drug addiction during the 12 months before the screening visit
* Active malignancy or history of malignancy in the 5 years prior to study entry
* Recent COVID-19 infection: within 60 days of recovery from infection
* Vaccination(s) within the last 60 days (including vaccines for SARS-CoV-2/COVID- 19)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes from baseline in physical examination | Baseline up to 5 years
  Safety and tolerability will be assessed by evaluating the number of patients with clinically significant changes from baseline in physical examination as assessed by an assessment of general appearance (head, eyes, ears, nose, and throat), as well as review of cardiovascular, dermatologic, gastrointestinal, genitourinary, lymphatic, musculoskeletal, neurologic and respiratory systems. Directed physical examinations at protocol-specified visits will be based on the patient's clinical status and will include general appearance, cardiovascular, gastrointestinal, neurologic, and respiratory assessments. Clinically significant changes from baseline will be captured as AEs.
Number of patients with clinically significant changes in vital signs from baseline | Baseline up to 5 years
  Safety and tolerability will be assessed by evaluating the number of patients with clinically significant changes from baseline in vital signs, including temperature, respiratory rate, seated blood pressure, and pulse.
Number of patients with clinically significant changes in total (IgG) IDUA antibody titres from baseline | Baseline up to 5 years
  Safety and tolerability will be assessed by evaluating the number of patients with clinically significant changes from baseline in total (IgG) antibody titres against IDUA
Number of patients with clinically significant changes in clinical laboratory tests from baseline | Baseline up to 5 years
  Safety and tolerability will be assessed by evaluating the number of patients with clinically significant changes from baseline in clinical laboratory tests, including hematology, serum chemistry, and urinalysis.
Number of patients with clinically significant changes in treatment-emergent adverse events (TEAE) from baseline, as assessed by CTCAE v5.0. | Baseline up to 5 years
  Safety and tolerability will be assessed by evaluating the number of patients with clinically significant changes from baseline in TEAEs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
To evaluate and Characterize effect of SIG-005 in levels of α-L-iduronidase (IDUA) in blood after administration of SIG-005 | Baseline up to 5 years
  To evaluate and characterize levels of IDUA and leukocyte count in blood plasma from time of baseline up to 5 years post-administration of SIG-005.
To evaluate and Characterize effect of SIG-005 on glycosaminoglycans (GAG) levels in urine following administration of SIG-005. | Baseline up to 5 years
  Total GAG, HS and DS levels in urine and any clinically significant changes will be assessed from time of baseline up to 5 years post-administration of SIG-005.
To evaluate and Characterize effect of SIG-005 MRI images of liver and spleen volume | Baseline up to 5 years
  Non-contrast MRI of the liver and spleen will be performed to determine any clinically significant changes in liver or spleen volume from time of baseline up to 5 years post-administration of SIG-005.
To evaluate and Characterize effect of SIG-005 on cardiac measurements via electrocardiogram (ECG) | Baseline up to 5 years
  Resting 12-lead ECG assessments will be performed to determine any clinically significant changes in cardiac measurements from time of baseline up to 5 years post-administration of SIG-005.

OTHER OUTCOMES:
To assess the effect of SIG-005 on health assessment and health-related quality of life | Baseline up to 5 years
  The effect of SIG-005 on health and health-related quality of life will be measured as changes from baseline in responses to the 12-Item Short Form Health Survey (SF-12) and the 5-level EuroQuol EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Clinical Study Site, Porto Alegre, Brazil
- United Kingdom (2):
  - Clinical Study Site, London
  - Clinical Study Site, Salford

IPD SHARING:
Plan to Share IPD: Undecided